CLINICAL TRIAL: NCT07058363
Title: Effects of Progressive Relaxation Exercises Applied to Patients With Ankylosing Spondylitis on Pain and Fatigue Levels
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Hilal BENZER, Principal Investigator, University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GaziantepU
Record Dates: First submitted 2025-05-28; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Ankylosing Spondylitis
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Intervention Model Description: This study was planned as a randomized, controlled and experimental study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PGE İntervention (Experimental): PGE will be applied to the patients in the PGE group by the assistant researcher in the first session using a one-on-one and face-to-face interview technique, approximately 20-25 minutes. Then, PGE application will be continued with online interviews to be conducted by the assistant researcher three days a week in the mornings for eight weeks. Pain levels of patients who receive PGE will be assessed with VAS after each session and the results will be compared with the control group that does not receive PGE. In addition, fatigue levels of patients in the PGE group will be assessed with PYS every four weeks before PGE, in the 4th and 8th weeks. Fatigue levels of patients in the control group will be assessed with PYS every four weeks at the beginning, in the 4th and 8th weeks.
  Interventions: Other: Progressive Relaxation Exercises
- PGE Control (No Intervention): The fatigue levels of the control group will be assessed with the PMS every four weeks, at the beginning, week 4 and week 8. At the end of the study, if the patients in the control group wish, they will be taught progressive relaxation exercises and allowed to do them.

INTERVENTIONS:
Other: Progressive Relaxation Exercises — Progressive Relaxation Exercises are defined as "a method that provides relaxation throughout the body by voluntary, regular relaxation of large muscle groups in the human body." The main purpose of relaxation exercises is for individuals to feel the difference between tension and relaxation in the muscles and to learn to relax on their own in cases of tension.
  Arms: PGE İntervention

SUMMARY:
Ankylosing spondylitis (AS) is a chronic rheumatic disease with unique clinical, pathophysiological, radiographic and genetic features, the etiology of which is not known for sure, and is characterized by sacroiliac and spinal joint involvement. It is reported that this disease affects one in every 200 people, is usually diagnosed years after the onset of symptoms, and negatively affects quality of life. The prevalence of AS is between 0.2% and 1.1%, and symptoms begin before the age of 30 in approximately 80% of cases. The main complaints of patients diagnosed with AS include pain, joint stiffness, fatigue, and functional limitations of various degrees. Functional limitations resulting from inflammation and/or bone formations affect daily life activities, especially the person's ability to participate in leisure and domestic activities, and work productivity, and can limit social roles in the family and society. It is reported in the literature that regular PGE reduces pain and fatigue, facilitates the transition to sleep, and improves quality of life. In this context, this study aimed to evaluate the effect of PGE in reducing pain and fatigue frequently experienced by AS patients and to contribute to symptom management.

DETAILED DESCRIPTION:
1. Research Design/Model/Type:

   Method of the study: This study is planned as randomized, controlled and experimental. The universe of the study will consist of all patients who applied to the rheumatology clinic of Gaziantep University Şahinbey Research and Training Hospital, and the sample will consist of patients diagnosed with AS who meet the inclusion criteria according to the power analysis. Patients will be divided into control and PGE groups using a simple random sampling method. It has been determined that the duration/frequency of progressive relaxation exercises is not specific/standardized and the total number of sessions also varies, but PGE is mainly applied for 4-12 weeks, two or three sessions per week. Therefore, in this study, it is planned to apply PGE three times per week for eight weeks, a total of 24 sessions.

   Place and Time of the Study This study will be conducted in the Gaziantep University Şahinbey Research and Training Hospital Rheumatology polyclinic and clinic. The planned study period is 18 months after obtaining the necessary ethics committee and institutional permissions.
2. Study Group/Sample of the Study: In the power analysis, the study titled 'Effect of progressive relaxation exercises on pain perception and quality of life in pregnant women with low back pain' by Baykal (2008) was taken as reference; in order to find a statistically significant expectation that a large effect size (d=1.46) would occur between the 4th week VAS values of the intervention and control groups, the minimum number required in each group was determined as 11 (α=0.05; 1-β=0.90). In order for the intervention and control groups to be balanced, it was decided to include the same number of control groups. However, considering possible losses, it is aimed to include a minimum of 25 patients in each group. Power analysis was performed in Gpower 3.9.1 software.
3. Data Collection Tools to be Used in the Project/Research:

   1. Question Form: This form, prepared by the researchers after examining the relevant literature, consists of questions that question the gender, age, marital status, education level, diagnosis period, and medication use of the individuals.
   2. Visual Analog Scale (VAS): This scale is a measurement tool with 10 on one end and 0 on the other. The patient is asked to mark a point corresponding to the pain intensity they feel. They are told to accept the time they do not feel any pain as "0" and the time they feel the most severe pain as "10", and the numerical value found shows the patient's pain intensity. The pain levels of the group that will do progressive relaxation exercises will be evaluated with VAS after each PGE. In addition, the pain levels of the patients in the control group will be evaluated with VAS simultaneously with the group that receives PGE.
   3. Piper Fatigue Scale (PFS): It is a tool consisting of 22 items and four sub-dimensions that subjectively measure one-month fatigue. Each item is rated from weak (1 point) to strong (10 points). The total score is found by summing up the answers to all items and dividing by the number of items. The maximum score that can be obtained from the scale is 10, and the minimum score is 0. An increase in the score means that the fatigue felt by the person is high. The fatigue level of the patients in the group that will perform progressive relaxation exercise and the control group will be evaluated with the PFS every four weeks, at the beginning, the 4th week and the 8th week.

   Progressive Relaxation Exercise Application Process: Before starting the study, the patients will be informed by the researcher in a room allocated for the study in the outpatient clinic and their permissions will be obtained. Later, in the evaluation made with VAS, patients with pain scores above 0 will be randomised using a simple random number table, PGE and control groups will be randomised. The patients in the PGE group will be informed about the PGE prepared by the Turkish Psychologists Association in the first session by the assistant researcher, using a one-on-one and face-to-face interview technique, in approximately 20-25 minutes. In this interview, individuals will also be told how to tense and relax certain areas of the body and how to complete the session within the scope of PGE, and they will be enabled to do so. At the end of the first interview, the internet access of the patients in the PGE group will be checked, and the patients will be informed about the content of the online interview techniques. Then, for eight weeks, the PGE application will be continued with online interviews to be held by the assistant researcher three days a week and in the morning. Since the duration of PGE will be 20-25 minutes, patients will be divided into groups of five and for individuals who cannot participate in the PGE program planned to be implemented at the patients' homes, repeat sessions will be planned on the same day according to their availability and their participation will be ensured every day. The pain levels of patients who receive PGE will be assessed with VAS after each session and the results will be compared with the control group that did not receive PGE. In addition, the fatigue levels of patients in the PGE group will be assessed with PYE every four weeks, before PGE, in the 4th week and in the 8th week. The fatigue levels of the control group will be assessed with PYE every four weeks, at the beginning, in the 4th week and in the 8th week. At the end of the study, patients in the control group will be taught progressive relaxation exercises and will be allowed to do them if they wish.
4. Evaluation of Project/Research Data: Data will be evaluated using the Statistical Package for Social Sciences-SPSS 25.0 package program, and frequency, percentage, mean and standard deviation will be used as descriptive statistics, and Shapiro Wilk test will be used to check the normal distribution of continuous variables. Student t, Chi-square, Mann-Whitney U and Kruskal Wallis, Anova tests will be applied under appropriate conditions to examine the differences between categorical variables. The statistical significance level will be accepted as p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Having AS diagnosis
* Volunteering to participate in the study
* Being over 18 years of age
* Having internet access

Exclusion Criteria:

* Having an orthopedic disability that prevents PGE
* Being pregnant
* Scoring 24 or less from the Mini Mental Test for individuals over 65 years of age
* Wanting to leave the study
* Having any psychiatric problems
* Not using a communication tool that allows online interviews
* Scoring "0" for pain and fatigue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2026-07-15 (Estimated); Study Completion 2027-01-15 (Estimated)

PRIMARY OUTCOMES:
PGE intervention and control | 8 weeks later
  When comparing the results of the PGE(PRE) Intervention and Control Group; A comparison will be made as to whether the applied Progressive Relaxation Exercises have an effect on pain and fatigue or not.
  Data will be evaluated using the Statistical Package for Social Sciences-SPSS 25.0 package program, and frequency, percentage, mean and standard deviation will be used as descriptive statistics, and Shapiro Wilk test will be used to check the normal distribution of continuous variables. Student t, Chi-square, Mann-Whitney U and Kruskal Wallis, Anova tests will be applied under appropriate conditions to examine the differences between categorical variables. The statistical significance level will be accepted as p<0.05.
VAS | 8 weeks later
  Visual Analog Scale (VAS): This scale is a measurement tool with 10 on one end and 0 on the other. The patient is asked to mark a point that corresponds to the intensity of pain they feel. They are told to accept the time they do not feel any pain as "0" and the time they feel the most severe pain as "10", and the numerical value found shows the patient's intensity of pain. The pain levels of the group that will do progressive relaxation exercises will be assessed with VAS after each PGE. In addition, the pain levels of the patients in the control group will be assessed with VAS simultaneously with the group that receives PGE.
PİPER | 0-4-8 weeks later
  Fatigue Piper Fatigue Scale (PFS): It is a tool consisting of 22 items and four sub-dimensions that subjectively measure one-month fatigue. Each item is rated from weak (1 point) to strong (10 points). The total score is found by summing up the answers to all items and dividing by the number of items. The maximum score that can be obtained from the scale is 10, and the minimum score is 0. An increase in the score means that the fatigue felt by the person is high. The fatigue level of the patients in the group that will do progressive relaxation exercises and the control group will be evaluated with the PFS every four weeks, at the beginning, the 4th week and the 8th week.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Ovayolu, Prof. Dr., Study Director — https://www.gaziantep.edu.tr/

IPD SHARING:
Plan to Share IPD: No
The research data will remain confidential by the researchers.